CLINICAL TRIAL: NCT03578536
Title: Effect of Constraint-Induced Gaming Therapy in an Acute Care Setting
Acronym: CIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2726-P; RX-002726-01A1 (Other Grant/Funding Number: VA-RR&D-SPIRE)
Record Dates: First submitted 2018-06-04; First posted 2018-07-06 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-04

CONDITIONS: Stroke
Keywords: Stroke; Therapy, Occupational; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Intervention Model Description: Single Group: Clinical trials with a single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CIT with Recovery Rapids (Experimental): This project will develop a therapeutic model that promotes use of the impaired arm and hand. Researchers often call this type of therapy "constraint induced therapy". In this study, participants focus on using the impaired limb rather than the unaffected limb. Study participants will only be able to play the game using the impaired limb.
  A small group of patients will participate in a question and answer session about preferences for activities which make up transfer tasks. Patients will also receive automated reminders to use the impaired arm throughout the day. Twelve (12) Veterans will be recruited annually from the inpatient Stroke Specialty Program. Six (6) patients will be assigned to the Treatment group and receive the intervention. The remaining six (6) will receive the current standard of care. Outcome measures will include motor function tests that evaluate upper extremity function.
  Interventions: Device: Recovery Rapids

INTERVENTIONS:
Device: Recovery Rapids — This project utilizes a new gaming system technology called Recovery Rapids. The game is custom-made by Games That Move You, LLC and runs on an XBOX platform with motion input via a Kinect system.

SUMMARY:
Current protocols for therapy on a rehabilitation unit call for intensive rehabilitation composed of high intensity, long duration therapy. Evidence from brain healing and animal research, along with motor learning principles suggest that a treatment program composed of short duration therapy sessions distributed throughout the day may provide better rehabilitation outcomes for stroke patients. Such a program can be implemented using constraint-induced therapy in which the Veteran is provided with opportunities to use the affected limb while participating in a video game and completing complementary tasks in therapy. Additionally, rehabilitation outcomes may improve if Veterans are provided with regular opportunities to participate in gaming therapy at home after discharge from the hospital rather than having to travel to a clinic or receive limited or no follow-up in rural areas.

This project will develop a therapeutic model that promotes use of the impaired arm and hand. Researchers often call this type of therapy "constraint induced therapy". In this study, participants focus on using the impaired limb rather than the unaffected limb. A small group of patients will participate in a question and answer session about preferences for activities which make up transfer tasks. Up to twenty-four (24) Veterans inpatient with hemiparesis due to stroke in the brain will be recruited from the Minneapolis VA Health Care System. Study participants will only be able to play the game using the impaired limb. Participants may also receive automated reminders to use the impaired arm throughout the day. Gaming will occur in patient room and during occupational therapy. Participants will have the option of being discharged with the gaming system for continued gameplay. Outcome measures will include motor function tests that evaluate upper extremity function.

DETAILED DESCRIPTION:
Research Question

The two questions to be answered by this study are: 1) To what extent does game-based CI therapy (with the Transfer Package) increase use of the more affected upper extremity from inpatient rehabilitation through subacute follow-up.

2) What is the clinical effectiveness of distributed gaming CI therapy for improving motor function of the more affected upper extremity at 3 months post-discharge.

Background

Constraint-Induced (CI) Movement therapy is arguably the best treatment paradigm to pilot throughout the continuum of care because it is established as the most empirically-supported intervention in subacute and chronic stroke and is more effective than standard care in acute stroke when lower duration/intensity protocols are utilized. CI therapy has strong evidence of increased effectiveness relative to standard care in the only positive definitively-powered upper extremity trial. A limitation of the acute CI therapy literature is that most studies omitted the most essential component of CI therapy: The Transfer Package of behavioral techniques that promotes carry-over of training to daily activities. In absence of the Transfer Package, everyday use of the weaker arm does not substantially improve and structural brain plasticity and quality of life gains are not realized. Early studies also show that any treatment advantage of CI therapy acutely is not maintained in follow-up, suggesting that maintenance therapy post-discharge is likely essential for altering the recovery trajectory.

Clinical Significance

This work will have a positive impact on the field of rehabilitation because it offers a solution to the main barriers of delivering distributed empirically-based treatment within an inpatient rehabilitation setting. By providing a paradigm for delivering distributed upper extremity practice, the product of this work has the potential to improve post-stroke health outcomes, lower-cost, and maintain the continuity of treatment from inpatient rehabilitation to community care.

Methods

The project will involve participatory action research methods to identify potential barriers to implementation of this new intervention within the VA and to refine the treatment approach to meet the needs of an inpatient population. A focus group will involve at least 3 patients who are currently on the inpatient rehabilitation unit (or recently discharged), their families, and occupational therapy/physical therapy (OT/PT)/recreational therapy staff. This meeting will serve to finalize the treatment protocol for this study. Areas that will be addressed will include the "dosing" schedule for the game-based intervention and needed adaptations to the CI therapy Transfer Package techniques (described below) to promote maximal carry-over from trained activities to everyday use of the weaker upper extremity. Any needed modifications to the technology platform (e.g. data storage) will also be made to comply with the VA's regulatory policies regarding adoption of new technology.

Up to 24 stroke survivors with upper extremity hemiparesis will be enrolled. Participants have the option of taking the gaming system home after discharge.

Gaming CI Therapy (Approximate Schedule)

1. 30 total inpatient hours OT/PT:

   * One 30-minute session to teach game play
   * 4.5 hours devoted to Transfer Package
   * Remainder time spent in usual care activities
2. 14 hours independent game play while inpatient
3. 18 hours independent game play following discharge (30 min, 3 times weekly) over and above standard care (will be documented as covariate)
4. Optional use of smart watch with biofeedback

This study will be conducted at the Minneapolis Veterans Affairs Medical Center (MVAMC). The MVAMC is home to the Stroke Specialty Program (SSP), a Commission on Accreditation of Rehabilitation Facilities (CARF) accredited program. The SSP tailors rehabilitation for survivors of any stroke mechanism (hemorrhagic, occlusive, etc.) affecting any part of the brain. Services can be adapted for survivors with cognitive challenges. The SSP has averaged 41 admissions in the past three years, though 2017 has projected admissions over 50. Retrospective chart review demonstrates the primary diagnosis resulting from stroke to be hemiplegia in approximately half of the admissions. Most patients (85%) are older than 60 years, predominantly Caucasian (85%) or African-American (10%) and male (98%).

Study participants will be patients enrolled in the MVAMC Stroke Specialty Program. Prospective participants will be screened by study staff. A retrospective chart review will be conducted to review outcomes of patients who underwent stroke rehabilitation at the Minneapolis VA but did not receive the study intervention. These subjects will serve as a retrospective control.

ELIGIBILITY:
Inclusion Criteria:

* Veteran between 18 and 88 years of age
* Inpatient at the Minneapolis VAHCS
* Willing and able to give Informed Consent or meets criteria for surrogate consent
* Upper extremity hemiparesis resulting from stroke in the brain (including brainstem) or tumor resection at the discretion of the therapist
* Lives within vicinity of the Minneapolis VA

Exclusion Criteria:

* Complete loss of arm function
* No contact address or telephone
* Active substance use disorder or major uncontrolled psychiatric disorder

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H Hansen, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
There will be no sharing of the IPD. Only a de-identified data set will be available upon request from the PI.

REFERENCES:
- [Background] Morris DM, Uswatte G, Crago JE, Cook EW 3rd, Taub E. The reliability of the wolf motor function test for assessing upper extremity function after stroke. Arch Phys Med Rehabil. 2001 Jun;82(6):750-5. doi: 10.1053/apmr.2001.23183. PMID 11387578
- [Background] Taub E, Wolf SL. Constraint Induced Movement Techniques To Facilitate Upper Extremity Use in Stroke Patients. Top Stroke Rehabil. 1997 Jan;3(4):38-61. doi: 10.1080/10749357.1997.11754128. PMID 27620374

RESULTS

PARTICIPANT FLOW:
Groups:
- CIT With Recovery Rapids: This project will develop a therapeutic model that promotes use of the impaired arm and hand. Researchers often call this type of therapy "constraint induced therapy". In this study, participants focus on using the impaired limb rather than the unaffected limb. Study participants will only be able to play the game using the impaired limb.
  A small group of patients will participate in a question and answer session about preferences for activities which make up transfer tasks. Veterans will be recruited from the inpatient Stroke Specialty Program and be assigned to receive the intervention. Outcome measures will include motor function tests that evaluate upper extremity function.
  Recovery Rapids: This project utilizes a new gaming system technology called Recovery Rapids. The game is custom-made by Games That Move You, LLC and runs on an XBOX platform with motion input via a Kinect system.
Period: Overall Study
Arm/Group | CIT With Recovery Rapids
Started | 3
Completed | 2
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Veterans with stroke
Arm/Group | CIT With Recovery Rapids
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Action Research Arm Test (ARAT) [Mean (Full Range); unit: units on a scale] — ARAT scores range from 0-57 points, with 57 points indicating no upper extremity impairment, and 0 points indicating no upper extremity movement.
  units on a scale | 36 [32 to 38]

OUTCOME MEASURES:

1. Primary Outcome: Action Research Arm Test (ARAT)
Description: The ARAT is a 19-item observational method used to assess upper extremity function on four subscales (grasp, pinch, gross movement, and grip). ARAT scores range from 0-57 points, with 57 points indicating no upper extremity impairment, and 0 points indicating no upper extremity movement.
Time Frame: The ARAT was administered by OT at Day 0 (Enrollment), and discharge at 6 weeks post-enrollment for subject 1 and at 4 weeks post-enrollment for subject 2
Population: Veterans with stroke and impaired upper extremity function
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | CIT With Recovery Rapids
Number analyzed (Participants) | 2
units on a scale
  Baseline ARAT | 37.5 [37 to 38]
  Discharge ARAT | 47 [42 to 52]

2. Primary Outcome: Motor Activity Log (MAL) Change (Discharge MAL - Enrollment MAL)
Description: The Motor Activity Log (MAL) is a motivational tool to assist stroke survivors in identifying goal movements and tracking progress. The Quality of Movement (QOM) subscale has participants rate themselves on how well they perform various activities of daily living with their more affected arm on a 0-5 scale. Scores are averaged across items and range from 0-5, with higher scores indicating the participant's ability to use their affected arm just as well as before their stroke.
Time Frame: Performed at Day 0 (enrollment) and at discharge (at 6 weeks post-enrollment for subject 1 and 4 weeks post-enrollment for subject 2)
Population: Veterans with stroke and impaired upper extremity function.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | CIT With Recovery Rapids
Number analyzed (Participants) | 2
units on a scale | 2.7 [2.42 to 3]

3. Secondary Outcome: Wolf Motor Function Test (WMFT)
Description: The Wolf Motor Function Test (WMFT) is a time-limited method to evaluate upper extremity performance while providing insight into joint-specific and total limb movements.
Time Frame: The WMFT may be administered by OT at at Day 0 (Enrollment), discharge, and potentially at 3 months post-discharge.
Population: Veterans with stroke and impaired upper extremity function. Participants were room bound due to COVID and there was not enough space in their rooms to perform the assessment.
Arm/Group | CIT With Recovery Rapids
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of enrollment in the study until the end of study participation, an average of 1 month.
Description: Did not differ from clinicaltrials.gov definitions.
Arm/Group | CIT With Recovery Rapids
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
The majority of Veterans approached for our study had nearly full day-time schedules limiting recruitment. We also experienced major problems related to the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT03578536/Prot_SAP_000.pdf